CLINICAL TRIAL: NCT02828358
Title: A Groupwide Pilot Study to Test the Tolerability and Biologic Activity of the Addition of Azacitidine (IND# 133688, NSC# 102816) to Chemotherapy in Infants With Acute Lymphoblastic Leukemia (ALL) and KMT2A(MLL) Gene Rearrangement
Brief Title: Azacitidine and Combination Chemotherapy in Treating Infants With Acute Lymphoblastic Leukemia and KMT2A Gene Rearrangement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-00973; NCI-2016-00973 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); s17-00488; AALL15P1 (Other: Children's Oncology Group); AALL15P1 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2016-07-07; First posted 2016-07-11 (Estimated); Results first posted 2021-10-26 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-01

CONDITIONS: Acute Leukemia of Ambiguous Lineage; B Acute Lymphoblastic Leukemia; Mixed Phenotype Acute Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Burkitt Lymphoma | interventions — Azacitidine; Specimen Handling; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Hydrocortisone; hydrocortisone hemisuccinate; Leucovorin; Magnetic Resonance Spectroscopy; Mercaptopurine; azathiopurine; Methotrexate; merphos; pegaspargase; Prednisolone; Methylprednisolone; Thioguanine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (azacitidine, combination chemotherapy) (Experimental): See Detailed Description
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Procedure: Echocardiography; Drug: Hydrocortisone Sodium Succinate; Drug: Leucovorin; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Pegaspargase; Drug: Prednisolone; Drug: Thioguanine; Drug: Vincristine; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Azacitidine — Given IV
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Cytarabine — Given IV, SC, IT
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin — Given IV
  Other Names: Daunomycin; Daunorrubicina; DNR; Leukaemomycin C; Rubidomycin; Rubomycin C
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Dexamethasone — Given PO, NG, IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Drug: Hydrocortisone Sodium Succinate — Given IT
  Other Names: (11beta)-21-(3-Carboxy-1-oxopropyl)-11,17-dihydroxypregn-4-ene-3,20-dione, Monosodium Salt; A-Hydrocort; Buccalsone; Corlan; Cortisol Sodium Succinate; Cortop; Efcortelan; Emergent-EZ; Flebocortid; Hidroc Clora; Hycorace; Hydro-Adreson; Hydrocort; Hydrocortisone 21-Sodium Succinate; Hydrocortisone Na Succinate; Kinogen; Nordicort; Nositrol; Sinsurrene; Sodium hydrocortisone succinate; Solu-Cortef; Solu-Glyc
Drug: Leucovorin — Given PO, IV
  Other Names: Folinic acid
Drug: Leucovorin Calcium — Given PO, IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Mercaptopurine — Given PO, NG
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IT, IV, PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Pegaspargase — Given IV
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Drug: Prednisolone — Given PO, NG
  Other Names: (11beta)-11,17,21-Trihydroxypregna-1,4-diene-3,20-dione; .delta.1-Hydrocortisone; Adnisolone; Aprednislon; Capsoid; Cortalone; Cortisolone; Dacortin H; Decaprednil; Decortin H; Delta(1)Hydrocortisone; Delta- Cortef; Delta-Cortef; Delta-Diona; Delta-F; Delta-Phoricol; Delta1-dehydro-hydrocortisone; Deltacortril; Deltahydrocortisone; Deltasolone; Deltidrosol; Dhasolone; Di-Adreson-F; Dontisolon D; Estilsona; Fisopred; Frisolona; Gupisone; Hostacortin H; Hydeltra; Hydeltrasol; Klismacort; Kuhlprednon; Lenisolone; Lepi-Cortinolo; Linola-H N; Linola-H-Fett N; Longiprednil; Metacortandralone; Meti Derm; Meticortelone; Opredsone; Panafcortelone; Precortisyl; Pred-Clysma; Predeltilone; Predni-Coelin; Predni-Helvacort; Prednicortelone; Prednisolonum; Prelone; Prenilone; Sterane
Drug: Thioguanine — Given PO, NG
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This pilot phase II trial studies the side effects of azacitidine and combination chemotherapy in infants with acute lymphoblastic leukemia and KMT2A gene rearrangement. Drugs used in chemotherapy, such as methotrexate, prednisolone, daunorubicin hydrochloride, cytarabine, dexamethasone, vincristine sulfate, pegaspargase, hydrocortisone sodium succinate, azacitidine, cyclophosphamide, mercaptopurine, leucovorin calcium, and thioguanine work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the tolerability of azacitidine in addition to Interfant-06 standard chemotherapy in infants with newly diagnosed acute lymphoblastic leukemia (ALL) with KMT2A gene rearrangement (KMT2A-R).

SECONDARY OBJECTIVE:

I. To evaluate the biologic activity of azacitidine by pharmacodynamic assessment of global deoxyribonucleic acid (DNA) methylation in peripheral blood mononuclear cells (PBMCs) of infants treated with azacitidine.

EXPLORATORY OBJECTIVES:

I. To determine the 5 year event-free survival (EFS) of infants with KMT2A-R treated with azacitidine in addition to Interfant-06 standard chemotherapy.

II. To correlate minimal residual disease (MRD) with outcome in the context of the protocol therapy.

III. To perform pharmacokinetic (PK) testing of azacitidine in infants. IV. To test the expansion of infant T lymphocytes by stimulation with artificial antigen presenting cells identical to those used in chimeric antigen receptor T-cell (CART)-19 production.

V. To collect pharmacodynamic (PD) data for asparaginase activity following pegaspargase administration in infants.

OUTLINE:

INDUCTION CHEMOTHERAPY: Patients receive methotrexate intrathecally (IT) on days 1 and 29, prednisolone orally (PO) or nasogastrically (NG) three times daily (TID) on days 1-7, daunorubicin hydrochloride intravenously (IV) over 1-15 minutes on days 8-9, cytarabine IV over 30 minutes on days 8-21 and IT on day 15, dexamethasone PO, NG, or IV TID on days 8-28, vincristine sulfate IV over 1 minute on days 8, 15, 22, and 29, pegaspargase IV over 1-2 hours or intramuscularly (IM) on day 12, and hydrocortisone sodium succinate IT on days 15 and 29 in the absence of disease progression or unacceptable toxicity. Only patients with KMT2A-R continue to post-induction chemotherapy.

POST-INDUCTION CHEMOTHERAPY:

AZACITIDINE BLOCK I: Prior to CONSOLIDATION, patients receive azacitidine IV over 10-40 minutes daily for 5 days in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Following completion of AZACITIDINE BLOCK I, patients receive cyclophosphamide IV over 30-60 minutes on days 1 and 29, mercaptopurine PO or NG daily on days 1-28, cytarabine IV or subcutaneously (SC) daily on days 3-6, 10-13, 17-20, and 24-27 and IT on day 10, methotrexate IT on day 24, and hydrocortisone sodium succinate IT on days 10 and 24 in the absence of disease progression or unacceptable toxicity.

AZACITIDINE BLOCK II: Prior to INTERIM MAINTENANCE, patients receive azacitidine as in AZACITIDINE BLOCK I

INTERIM MAINTENANCE: Following completion of AZACITIDINE BLOCK II, patients receive mercaptopurine PO or NG daily on days 1-14, methotrexate IV over 24 hours on days 1 and 8 and IT on days 2 and 9, leucovorin calcium PO or IV on days 3-4 and 10-11, hydrocortisone sodium succinate IT on days 2 and 9, cytarabine IV over 3 hours every 12 hours on days 15-16 and 22-23 for a total of 8 doses, and pegaspargase IV over 1-2 hours or IM on day 23 in the absence of disease progression or unacceptable toxicity.

AZACITIDINE BLOCK III: Prior to DELAYED INTENSIFICATION PART I, patients receive azacitidine as in AZACITIDINE BLOCK I.

DELAYED INTENSIFICATION PART I: Following completion of AZACITIDINE BLOCK III, patients receive pegaspargase IV over 1-2 hours or IM on day 1, dexamethasone PO, NG, or IV TID on days 1-14 and 15-21 with a taper on days 15-21, thioguanine PO or NG daily on days 1-28, vincristine sulfate IV over 1 minute on days 1, 8, 15, and 22, daunorubicin hydrochloride IV over 1-15 minutes on days 1, 8, 15, and 22, cytarabine IV or SC on days 2-5, 9-12, 16-19, and 23-26 and IT on days 1 and 15, and hydrocortisone sodium succinate IT on days 1 and 15 in the absence of disease progression or unacceptable toxicity.

AZACITIDINE BLOCK IV: Prior to DELAYED INTENSIFICATION PART II, patients receive azacitidine as in AZACITIDINE BLOCK I.

DELAYED INTENSIFICATION PART II: Following completion of AZACITIDINE BLOCK IV, patients receive thioguanine PO or NG daily on days 1-14, cyclophosphamide IV over 15-30 minutes on days 1 and 15, cytarabine IV or SC on days 2-5 and 9-12 in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Following DELAYED INTENSIFICATION PART II, patients receive mercaptopurine PO or NG on days 1-168, methotrexate IT on day 1 and 92 and PO once weekly on days 8-91 and 98-168, hydrocortisone sodium succinate IT on day 1, 57, and 99, and cytarabine IT on day 57. Starting on day 169, patients receive mercaptopurine PO or NG on days 1-84 and methotrexate PO once weekly. Cycles repeat every 84 days for 2 years from the start of INDUCTION CHEMOTHERAPY in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo collection of blood sample and an echocardiogram (ECHO) or multigated acquisition (MUGA) scan on study. Patients may also undergo computed tomography (CT) or magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Infants must be > 36 weeks gestational age at the time of enrollment
* Patients must have newly diagnosed B lymphoblastic leukemia (2008 World Health Organization [WHO] classification) (also termed B-precursor acute lymphoblastic leukemia) or acute leukemia of ambiguous lineage (ALUL), which includes mixed phenotype acute leukemia (MPAL); for patients with ALUL, the morphology and immunophenotype must be at least 50% B lymphoblastic
* Central nervous system (CNS) status must be determined based on a sample obtained prior to the administration of any systemic or intrathecal chemotherapy, with the exception of steroid pretreatment

Exclusion Criteria:

* Patients with known absence of KMT2A-rearrangement leukemia prior to enrollment
* Patients with Down syndrome
* Patients with secondary B acute lymphoblastic leukemia (B-ALL) that developed after treatment of a prior malignancy with cytotoxic chemotherapy
* With the exception of steroid pretreatment or the administration of intrathecal methotrexate or intrathecal cytarabine, receipt of any other prior cytotoxic chemotherapy for either the current diagnosis of B-ALL or any cancer diagnosed prior to the initiation of protocol therapy on AALL15P1

Max Age: 364 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rishi S Kotecha, Principal Investigator — Children's Oncology Group
Locations (170):
- United States (157):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- Canada (8):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
- Puerto Rico (3):
  - HIMA San Pablo Oncologic Hospital, Caguas
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Guest EM, Kairalla JA, Devidas M, Hibbitts E, Carroll AJ, Heerema NA, Kubaney HR, August MA, Ramesh S, Yoo B, Farooqi MS, Pauly MG, Wechsler DS, Miles RR, Reid JM, Kihei CD, Gore L, Raetz EA, Hunger SP, Loh ML, Brown PA. Azacitidine as epigenetic priming for chemotherapy is safe and well-tolerated in infants with newly diagnosed KMT2A-rearranged acute lymphoblastic leukemia: Children's Oncology Group trial AALL15P1. Haematologica. 2024 Dec 1;109(12):3918-3927. doi: 10.3324/haematol.2024.285158. PMID 38867582

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants less than 1 year of age with newly diagnosed B lymphoblastic leukemia (also termed B-precursor acute lymphoblastic leukemia) or acute leukemia of ambiguous lineage
Pre-assignment Details: Enrolled patients receive common induction therapy. Genetic evaluation results in patients being stratified into KMT2A-Germline and KMT2A-Rearranged groups. KMT2A-Germline patients go off protocol therapy post-induction.
Groups:
- KMT2A-Rearranged: INDUCTION: Same as KMT2A-Germline (Group 2). AZACITIDINE (AZA) I: AZA over 10-40 minutes for 5 days. CONSOLIDATION: cyclophosphamide days 1/29; mercaptopurine (6-MP) days 1-28; ARA-C days 3-6, 10-13, 17-20, 24-27; MTX IT day 24; HC days 10/24. AZA II: Same as AZA I. INTERIM MAINTENANCE: 6-MP days 1-14; MTX 1/2/8/9; leucovorin calcium days 3-4,10-11; HC days 2/9; ARA-C days 15-16, 22-23; PEG day 23. AZA III: Same as AZA I. DELAYED INTENSIFICATION (DI) I: PEG day 1; dexamethasone days 1-14, 15-21; thioguanine days 1-28; vincristine sulfate and daunorubicin hydrochloride days 1/8/15/22; ARA-C days 1-5, 9-12, 15-19, 23-26; HC on days 1/15. AZA IV: Same as AZA I. DI II: thioguanine days 1-14; cyclophosphamide days 1/15; ARA-C days 2-5, 9-12. MAINTENANCE: 6-MP days 1-168, MTX IT day 1/92; MTX weekly days 8-91,98-168; HC day 1/57/99; ARA-C day 57. Starting day 169, 6-MP days 1-84 and MTX weekly. Cycles repeat every 84 days for 2 years from start of Induction.
- KMT2A-Germline: Induction: Methotrexate intrathecally (IT) on days 1 and 29, prednisolone orally (PO) or nasogastrically (NG) three times daily (TID) on days 1-7, daunorubicin hydrochloride intravenously (IV) over 1-15 minutes on days 8-9, cytarabine (ARA-C) IV over 30 minutes on days 8-21 and IT on day 15, dexamethasone PO, NG, or IV TID on days 8-28, vincristine sulfate IV over 1 minute on days 8, 15, 22, and 29, pegaspargase (PEG) IV over 1-2 hours or intramuscularly (IM) on day 12, and hydrocortisone sodium succinate (HC) IT on days 15 and 29 in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | KMT2A-Rearranged | KMT2A-Germline
Started | 56 | 22
Completed | 11 | 0
Not Completed | 45 | 22
Not completed — Physician Decision | 7 | 1
Not completed — Treatment Failure | 6 | 0
Not completed — Patients without KMT2A rearrangement | 0 | 21
Not completed — Refusal of further protocol therapy | 2 | 0
Not completed — Relapse | 25 | 0
Not completed — Still on therapy | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KMT2A-Rearranged | KMT2A-Germline | Total
Number analyzed (Participants) | 56 | 22 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 56 | 22 | 78
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 0.48 (0.29) | 0.74 (0.2) | 0.55 (0.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 12 | 47
  Male | 21 | 10 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 4 | 15
  Not Hispanic or Latino | 40 | 17 | 57
  Unknown or Not Reported | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 40 | 15 | 55
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 9 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of Azacitidine in Combination With Interfant-06 Standard Chemotherapy in Evaluable Infant Patients With Newly Diagnosed ALL With KMT2A Gene Rearrangement (KMT2A-R). KMT2A Gene Rearrangement (KMT2A-R)
Description: Proportion of KMT2A-Rearranged patients treated with azacitidine with Dose Limiting Toxicities (DLTs) from the first course of azacitidine administration up to fourth course of azacitidine administration.
Time Frame: 6 months
Population: KMT2A-Rearranged patients evaluable for dose-limiting toxicity assessment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | KMT2A-Rearranged
Number analyzed (Participants) | 31
percentage of participants | 6.45 [0 to 15.10]

2. Secondary Outcome: Biologic Activity, Defined as Global Deoxyribonucleic Acid (DNA) Methylation Change in Peripheral Blood Mononuclear Cells (PBMC)s; Day 1 Prior to First Course of Azacitidine
Description: Will calculate the percentage of CpG site methylation for all patients before the first course of azacitidine. Mean and standard deviation will be reported.
Time Frame: Week 6, Day 1 (Following the induction phase (35 days), the first course of Azacitidine began around Week 6 of therapy)
Population: Patients with methylation data. KMT2A-Germline patients did not have data collected as they came off therapy at the end of Induction
Measure: Mean (Standard Deviation); unit: Percentage of CpG methylation
Arm/Group | KMT2A-Rearranged
Number analyzed (Participants) | 31
Percentage of CpG methylation | 78.17 (1.62)

3. Secondary Outcome: Biologic Activity, Defined as Global Deoxyribonucleic Acid (DNA) Methylation Change in Peripheral Blood Mononuclear Cells (PBMC)s; Day 5 of First Course of Azacitidine
Description: Will calculate the percentage of CpG site methylation for all patients after the first course of azacitidine. Mean and standard deviation will be reported.
Time Frame: Week 6, Day 5 (Following the induction phase (35 days), the first course of Azacitidine began around Week 6 of therapy)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of CpG methylation
Arm/Group | KMT2A-Rearranged
Number analyzed (Participants) | 31
Percentage of CpG methylation | 75.54 (2.68)

4. Secondary Outcome: Biologic Activity, Defined as Global Deoxyribonucleic Acid (DNA) Methylation Change in Peripheral Blood Mononuclear Cells (PBMC)s; Day 1 Prior to Second Course of Azacitidine
Description: Will calculate the percentage of CpG site methylation for all patients before the second course of azacitidine. Mean and standard deviation will be reported.
Time Frame: Week 13, Day 1 (Following induction phase (5 weeks), the first course of Azacitidine (1 week), and consolidation (6 weeks), the second course of Azacitidine began around Week 13 of therapy)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of CpG methylation
Arm/Group | KMT2A-Rearranged
Number analyzed (Participants) | 26
Percentage of CpG methylation | 76.5 (2.68)

5. Secondary Outcome: Biologic Activity, Defined as Global Deoxyribonucleic Acid (DNA) Methylation Change in Peripheral Blood Mononuclear Cells (PBMC)s; Day 5 of Second Course of Azacitidine
Description: Will calculate the percentage of CpG site methylation for all patients after the second course of azacitidine. Mean and standard deviation will be reported.
Time Frame: Week 13, Day 5 (Following induction phase (5 weeks), the first course of Azacitidine (1 week), and consolidation (6 weeks), the second course of Azacitidine began around Week 13 of therapy)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of CpG methylation
Arm/Group | KMT2A-Rearranged
Number analyzed (Participants) | 27
Percentage of CpG methylation | 74.52 (2.09)

6. Other Pre Specified Outcome: Event-free Survival (EFS)
Description: Five year EFS estimation will be calculated from time of enrollment. Standard errors and confidence intervals for EFS will be calculated using Peto's method.
Time Frame: Five years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Minimal Residual Disease (MRD)
Description: Descriptive analysis will be conducted to correlate MRD with the EFS for the KMT2A-R patients.
Time Frame: Five years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Pharmacokinetic (PK) Parameters of Azacitidine
Description: Pharmacokinetic (PK) testing and analysis of azacitidine in infants will be performed by Covance.
Time Frame: Two months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Expansion of Infant T Lymphocytes by Stimulation With Artificial Antigen Presenting Cells
Description: Optional biological study participation will explore the feasibility of T-cell collection for the purposes of chimeric antigen receptor (CAR) T-cell production from the peripheral blood in infants with ALL.
Time Frame: Three months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: PD Data for Asparaginase Activity Following Pegaspargase Administration
Description: Pharmacodynamic (PD) data for asparaginase activity following pegaspargase administration in infants will be collected, described, and correlated with EFS for the KMT2A-R patients.
Time Frame: Six months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | KMT2A-Rearranged | KMT2A-Germline
All-Cause Mortality (participants affected / at risk) | 17/56 | 1/22
Serious Adverse Events (participants affected / at risk) | 34/56 | 1/22
Other Adverse Events (participants affected / at risk) | 36/56 | 10/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KMT2A-Rearranged (N=56) | KMT2A-Germline (N=22)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 11 (11) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 5 (5) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0)
Rectal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KMT2A-Rearranged (N=56) | KMT2A-Germline (N=22)
Alanine aminotransferase increased (Investigations) | 4 (6) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (3) | 1 (1)
Catheter related infection (Infections and infestations) | 4 (4) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 17 (37) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 10 (10) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 6 (6) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 6 (8) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 4 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
GGT increased (Investigations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 3 (4) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Small intestine infection (Infections and infestations) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT02828358/Prot_SAP_000.pdf